CLINICAL TRIAL: NCT07384832
Title: Dynamic Stretching Versus Slider Neurodynamic Technique In Patients With Lumbar Radiculopathy
Brief Title: Comparative Effects Of Dynamic Stretching Versus Slider Neurodynamic Technique In Patients With Lumbar Radiculopathy
Acronym: DS vs SNT -LR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: University of Lahore Hospital (ULH) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0043
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Radiculopathy
Keywords: lumbar radiculopathy; sciatica
MeSH Terms: conditions — Radiculopathy; Sciatica | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study used a single-blind approach. This means that while the researchers knew which treatment each person was getting, the patients did not know if they were in the "Dynamic Stretching" group or the "Slider Neurodynamic" group. They were not told which exercise protocol was the main focus of the study or which one was expected to be more effective. This helps ensure that the patients' expectations did not influence the results or their reporting of pain levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Stretching + Routine Physiotherapy (Experimental): Participants in this group will receive Dynamic stretching Includes slump stretch, cat and camel, hamstring sweeps, child pose, and overhead lateral stretch.
  Protocol: 2 sets of 10-15 repetitions for 4 minutes with 1-minute rest intervals
  Interventions: Other: Dynamic stretching; Other: Routine physiotherapy
- Slider Neurodynamic Mobilization + Routine Physiotherapy (Active Comparator): Participants in this arm will receive Slider Neurodynamic Mobilization (NDM) along with routine physiotherapy. NDM slider techniques will be performed in the slump position according to a standardised protocol ( the patient to move actively and conversely from a position of neck and trunk flexion, knee flexion, and plantar flexion, to a position of neck and trunk extension, knee extension, and ankle dorsiflexion ) protocol: 3 sets of 1 minute slider movement with 1 minute rest interval
  Interventions: Other: slider neurodynamic mobilization; Other: Routine physiotherapy

INTERVENTIONS:
Other: Dynamic stretching — Dynamic stretching protocol will include:
  * Slump Stretch (4 minutes): The patient performed a slump stretch, seated with knees bent, extending one leg at a time while flexing the trunk forward to stretch the lumbar nerve roots.
  * Cat and Camel Stretch (4 minutes): The patient alternated between spinal flexion and extension while on hands and knees.
  * Hamstring Sweeps (4 minutes): The patient performed dynamic hamstring stretches, sweeping the leg forward and back to increase flexibility in the posterior chain.
  * Child's Pose Stretch (4 minutes): The patient performed a child's pose stretch to improve flexibility in the lower back and hips.
  * Overhead Lateral Stretch (4 minutes): The patient performed a side stretch to target the quadratus lumborum and obliques, releasing tension from the side of the back.
  Each dynamic stretch will be performed as follows:
  * 2 sets of 10-15 repetitions
  * 1-minute rest between sets
  * Performed 3 sessions/week for 6 weeks
  Arms: Dynamic Stretching + Routine Physiotherapy
Other: slider neurodynamic mobilization — Performed in the slump sitting position. Participants move from neck and trunk flexion with knee flexion and plantar flexion toward neck and trunk extension with knee extension and ankle dorsiflexion. The protocol consists of 3 sets of 1-minute slider movements, each followed by 1 minute of rest.
  Arms: Slider Neurodynamic Mobilization + Routine Physiotherapy
Other: Routine physiotherapy — 1. TENS : The patient was instructed to lie comfortably, and TENS was applied in conventional mode for 15 minutes at a frequency of 70 Hz and pulse width of 100 microseconds. Two 40x40 mm electrodes were placed on each side of the lumbosacral spine.
  2. Hot Moist Pack: A hot moist pack was applied to the lumbosacral and gluteal regions for 10 minutes in a prone position.
  3. Soft Tissue Mobilization: Soft tissue mobilization was performed for 5 minutes around the lumbar spine.
  4. Strengthening Exercises (5 minutes): Pelvic Tilt (2.5 minutes): The patient was instructed to lie on their back with knees bent and feet flat on the floor.
  Alternate Leg Extension (2.5 minutes): In the prone position, the patient lifted one leg for 10 seconds, lowered it, and then raised the other leg. Quads strengthening and adductor abductor strengthening was also done by using pillow and pressing the pillow.
  These exercises were performed for 2 sets of 15-20 reps with 1 minute rest interval

SUMMARY:
This study will be randomised clinical trial conducted at the University of Lahore Teaching Hospital, Lahore, Pakistan. A total of 72 participants will be selected and randomly allocated into two treatment groups (36 participants in each group) using the lottery method. All screened and willing participants who meet the eligibility criteria will be assigned to either Group A or Group B.

Group A will receive dynamic stretching along with routine physiotherapy. Routine physiotherapy will include TENS (15 minutes), hot moist pack (10 minutes), soft tissue mobilisation (5-7 minutes), abdominal bracing, pelvic tilt, and alternate leg extension exercises. The dynamic stretching part will include slump stretch, cat-camel stretch, hamstring sweeps, child pose stretch, and overhead lateral stretch. Each stretch will be performed in 2 sets of 15-20 repetitions with 1-minute rest between sets. Treatment will be provided four times per week for 6 weeks.

Group B will receive slider neurodynamic mobilisation along with the same routine phsiotherapy protocol as group A . Slider neurodynamic mobilisation will be performed in the slump position, sitting at the edge of the plinth with the thighs parallel to each other and arms crossing behind the back. The examiner asked the patient to move actively and conversely from a position of neck and trunk flexion, knee flexion, and plantar flexion, to a position of neck and trunk extension, knee extension, and ankle dorsiflexion with 3 sets of 1-minute sliders and 1-minute rest between sets. Treatment will be provided four times per week for 6 weeks.

All participants will undergo assessments at baseline, at the end of the 3rd week, and at the end of the 6th week.

DETAILED DESCRIPTION:
* Screening Participants who meet the inclusion criteria was recruited using a convenience sampling technique. This involves selecting participants who are readily available to participate in the study.
* Allocation Eligible participants was screened and informed about the study including its purpose, procedures, potential risks and benefits. Informed consent was obtained from each participant prior to their formal enrollment in the study.
* Randomization:

Following the baseline assessment, the randomization was conducted using the Online Randomizer tool (https://www.randomizer.org/). By specifying the group numbers, participants per group, and the total participants, unique identification numbers were generated for each participant.

• Blindness: This study a single blinded, the patients were kept blinded about the study and were not told related the exercise protocol they received.

• Intervention After taking consent, participants was selected based on the inclusion criteria. Sample of 72 was then be randomly divided into two groups.

All participants received a 35-minute treatment session, 4 days per week for 6 weeks, consisting of 15 minutes of routine physiotherapy and 20 minutes of a specific intervention:

Group A (Dynamic Stretching): Routine physiotherapy included TENS (70 Hz, 100 microseconds) for 15 minutes, hot moist packs for 10 minutes, and core strengthening (pelvic tilts and leg extensions). The main intervention was 20 minutes of dynamic stretching, including the slump stretch(The patient performed a slump stretch, seated with knees bent, extending one leg at a time while flexing the trunk forward to stretch the lumbar nerve roots), cat and camel(The patient alternated between spinal flexion and extension while on hands and knees.), hamstring sweeps(The patient performed dynamic hamstring stretches, sweeping the leg forward and back to increase flexibility in the posterior chain.), child's pose, and overhead lateral stretches(The patient performed a side stretch to target the quadratus lumborum and obliques, releasing tension from the side of the back.). Each exercise was performed For 4 minutes in 2 sets of 10-15 repetitions with 1 minute rest interval.

Group B (Slider Neurodynamic Technique): Routine physiotherapy matched Group A but included 5 minutes of soft tissue mobilization. The main intervention was the Slider Neurodynamic Mobilization (NDM). Patients were seated and performed rhythmic movements: moving from neck/trunk flexion and knee flexion to neck/trunk extension and knee extension. This movement is designed to "slide" the nerve through the spinal canal without over-tensioning it. This was performed in 3 sets of 1-minute intervals.

Clinical assessments for pain (NPRS), disability (MODI), and flexibility (MMST) were recorded at baseline, the 3rd week, and the 6th week to compare the efficacy of the two protocols.

ELIGIBILITY:
Inclusion Criteria:

* Both genders are included.
* Participants aged between 25 to 65 years.
* Symptoms that radiate below the buttocks, thigh/knee and lower leg for more than 4 weeks.
* Pain intensity (NPRS) >4/10
* Diagnosed with MRI to confirm any disc lesion.
* Had a positive slump test with reproduction of neurological symptoms and had functional disabilities in certain daily tasks, such as lifting or walking.

Exclusion Criteria:

* Patients with lumbar spondylolisthesis, pregnant women.
* Patients with ankylosing spondylitis, RA.
* Previous history of fracture or spinal laminectomy
* Systemic diseases like cardiovascular disease and metabolic diseases.
* Contraindication to exercises or usage of TENS.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (NPRS) | baseline, 3rd week, 6th week
  Pain Intensity will n=be measured using the numeric pain rating scale (NPRS) , where participants rate their pain on a scale from 0 to 10 (0= no pain, 10= worst possible pain). the scale will be used to assess changes in pain levels over the duration of the intervention.

SECONDARY OUTCOMES:
Functional Disability (Modified Oswestry Disability Index -MODI) | baseline,3rd week, 6th week
  Functional disability will be measured using the modified oswestry low back pain disability index, a validated questionnaire assessing limitations in everyday activities. scores range from 0-100 % with higher scores indicating greater disability. the measure will be used to determine changes in functional ability.
Lumbar Flexion Range of Motion (Modified-Modified Schober Test - MMST) | baseline, 3rd week, 6th week
  Lumbar flexion range of motion will be assessed using the Modified-Modified Schober Test (MMST). The test measures the change in distance between two points on the lumbar spine during forward flexion. Increased distance indicates improved lumbar mobility.

CONTACTS AND LOCATIONS:
Overall Officials: ASIM ARIF, PhD scholar, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaheen HM, Belgen Kaygisiz B. Comparison of different treatment positions of nerve slider technique for patients with low back pain: a randomized control trial. Eur J Phys Rehabil Med. 2025 Feb;61(1):82-92. doi: 10.23736/S1973-9087.24.08541-1. Epub 2025 Jan 28. PMID 39873676
- [Result] Nahid ZBS, Ahmed F, Islam MF, Rahman Z, Haque MF, Arju A, Islam MR, Moula G, Sarker B. Effectiveness of Shacklock's Neural Mobilization for Acute and Sub-Acute Lumbar Disc Prolapsed: A Randomized Controlled Trial. Health Sci Rep. 2025 May 26;8(5):e70872. doi: 10.1002/hsr2.70872. eCollection 2025 May. PMID 40432703
- [Result] de Ridder R, De Blaiser C, Verrelst R, De Saer R, Desmet A, Schuermans J. Neurodynamic sliders promote flexibility in tight hamstring syndrome. Eur J Sport Sci. 2020 Aug;20(7):973-980. doi: 10.1080/17461391.2019.1675770. Epub 2019 Oct 22. PMID 31578925
- [Result] Danazumi MS, Bello B, Yakasai AM, Kaka B. Two manual therapy techniques for management of lumbar radiculopathy: a randomized clinical trial. J Osteopath Med. 2021 Feb 26;121(4):391-400. doi: 10.1515/jom-2020-0261. PMID 33705612
- [Result] Ghaderi Niri H, Ghanavati T, Mostafaee N, Salahzadeh Z, Divandari A, Adigozali H, Ahadi J. Oswestry Disability Index, Roland-Morris Disability Questionnaire, and Quebec Back Pain Disability Scale: Responsiveness and Minimal Clinically Important Changes in Iranian People with Lumbar Disc Herniation Following Physiotherapy. Arch Bone Jt Surg. 2024;12(1):58-65. doi: 10.22038/ABJS.2023.72246.3366. PMID 38318303